CLINICAL TRIAL: NCT03642015
Title: The Effect of Music on Anxiety in Patients Prior to Gastrointestinal Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Yang Chia Chen, Principal Investigator, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TSGH-C97-151
Record Dates: First submitted 2018-08-14; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Music; Anxiety
Keywords: music; anxiety; digestive tract endoscopy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- listening music (Experimental): The participants in the music group selected the music they preferred from different genres. During the 15-min intervention period before the gastroscopy procedure, the experimental group rested by listening to music and sitting on a comfortable chair
  Interventions: Behavioral: Music listening
- Control (No Intervention): control group rested only by sitting on a comfortable chair

INTERVENTIONS:
Behavioral: Music listening — listening the music 15 min
  Arms: listening music

SUMMARY:
This study investigated the effect of listening to self-selected music on anxiety and physiological responses in patients prior to gastroscopy. A randomized controlled trial was conducted, in which patients scheduled for gastroscopy in a medical center located in Taipei, Taiwan, were enrolled. The experimental group listened to self-selected music with earphones for 15 min before the procedure, whereas the control group rested for 15 min. Blood pressure (BP), heart rate, respiratory rate, and anxiety level were measured immediately before and after the intervention.

DETAILED DESCRIPTION:
Potential study patients were referred from physicians. The research assistant described the study's purpose and procedure to the patients and explained their right to refuse or withdraw from the study without jeopardizing their procedure. In addition, the privacy of each patient's data was ensured by storing the data in a file that required a password to access. Personal identification was by no means included in the data file. In addition, the participants were assured that their data would not be used for purposes other than this research.

After obtaining their consent, the participants were randomly assigned into the music group or the control group by drawing lots. We brought the participants to a separate and quiet room in the waiting area to prevent environmental interference. First, the participants completed the study questionnaire; then, the research investigator measured their physiological parameters. The participants in the music group selected the music they preferred from different genres, namely Chinese pop, Taiwanese songs, western classical , light music, western pop, and nostalgic music. If a participant had no particular preference, music with a low tone, regular rhythm (approximately 60-80 beats per minute), and soft melody (light music, 5%) was used, as recommended by a previous study. During the 15-min intervention period before the gastroscopy procedure, the experimental group rested by listening to music and sitting on a comfortable chair, whereas the control group rested only by sitting on a comfortable chair. After the 15-min intervention, the patients' anxiety and physiological parameters were reassessed.

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age or older
* able to respond to questionnaires in Chinese. were excluded from the study.

Exclusion Criteria:

* with hearing loss who did not wear hearing aids
* patients who were unable to communicate verbally
* patients diagnosed with dementia, mental illness defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, or cognitive impairment

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-07-01 (Actual); Primary Completion 2008-09-01 (Actual); Study Completion 2009-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Anxiety after intervention immediately | baseline, 15 minute
  Anxiety was measured using the Chinese version of the 20-item State-Trait Anxiety Inventory-State Anxiety Scale (STAI-S), which demonstrated high reliability (Cronbach's alpha of 0.91) in patients with anxiety disorders.32 Total scores for state anxiety ranged from 20 to 80; higher scores indicated higher levels of anxiety.

SECONDARY OUTCOMES:
Change from Baseline Blood pressure after intervention immediately | baseline, 15 minute
  Blood Pressure was measured using a calibrated sphygmomanometer with an appropriately sized cuff.
Change from Baseline Heart Rate after intervention immediately | baseline, 15 minute
  Heart rate was measured through 1-min radial artery pulse counting.
Change from Baseline Respiratory Rate after intervention immediately | baseline, 15 minute
  Respiratory rate was determined by counting the number of breaths per minute during quiet breathing.